CLINICAL TRIAL: NCT04924595
Title: The Effect of a Personalised Training Programme on the Functional Ability and the Quality of Life of Candidates for Liver Transplantation
Brief Title: Exercise Intervention in Liver Transplant Candidates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Ilias Marios Oikonomou, Scientific Associate for the Surgical Department of Transplantation A.U.Th., Postgraduate Student, Medical Doctor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AUTh65/2021
Record Dates: First submitted 2021-05-30; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular treatment (No Intervention)
- Exercise Intervention (Experimental)
  Interventions: Behavioral: Personalised exercise

INTERVENTIONS:
Behavioral: Personalised exercise — Personalised exercise intervention including aerobic and resistance training
  Arms: Exercise Intervention

SUMMARY:
The aim of the study is to investigate the effect of personalised exercise interventions in liver transplant candidates, aiming to prevent or limit sarcopenia and frailty, as well as improving their cardiorespiratory health.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant candidates, accepted in the waiting list of the Surgical Department of Transplantation A.U.Th., General Hospital of Thessaloniki "Ippokratio".

Exclusion Criteria:

* Recent (<12 months) Acute Myocardial Infraction
* Recent (<12 months) brain strokes
* Uncontrolled and/or untreated arrythmia
* Hepatic encephalopathy
* Bed-bound patient
* Liver Transplantation
* Death

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-25 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline "Liver Frailty Index" value at 12 weeks | After 12-week exercise intervention
  A frailty index for patients with cirrhosis, comprised of three performance-based metrics
Change from Baseline "6 Minute Walking Test" value at 12 weeks | After 12-week exercise intervention
  A walking test for patients to evaluate their functional capacity

SECONDARY OUTCOMES:
VO2max | Before intervention initiation and after 12-week exercise intervention
  Maximum oxygen consumption during incremental exercise

CONTACTS AND LOCATIONS:
Overall Officials: Ilias M Oikonomou, MD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (2):
- Greece (2):
  - Laboratory of Sports Medicine, Thermi, Thessaloniki
  - Surgical Department of Transplantation A.U.Th., Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided